CLINICAL TRIAL: NCT01775865
Title: Targeting Inflammation to Treat Cardiovascular Aging in Humans (TIVA Study)
Brief Title: Targeting Inflammation to Treat Cardiovascular Aging
Acronym: TIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary L. Pierce (Other)
Responsible Party: Sponsor-Investigator, Gary L. Pierce, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201201739
Record Dates: First submitted 2013-01-04; First posted 2013-01-25 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-04

CONDITIONS: Vascular Stiffness; Endothelial Dysfunction; Diastolic Dysfunction
Keywords: aortic stiffness; endothelium-dependent dilation; vascular aging; oxidative stress; inflammation; nitric oxide; nuclear factor kappa B
MeSH Terms: conditions — Inflammation | interventions — salicylsalicylic acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Salsalate (Experimental): Salsalate capsule 1.5 g/day twice per day by mouth for 4 weeks
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): Placebo capsule twice per day by mouth for 4 weeks
  Interventions: Drug: Placebo (for salsalate)
- Young Control (No Intervention): No intervention; Baseline measurements only

INTERVENTIONS:
Drug: Salsalate — 4 weeks of daily salsalate
  Other Names: Disalcid; Mono-Gesic; Salflex; Salsitab
  Arms: Salsalate
Drug: Placebo (for salsalate) — 4 week of daily placebo
  Other Names: Placebo capsule sugar pill to mimic salsalate
  Arms: Placebo

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in the United States with older age being a primary risk factor. The number of adults greater than age 65 years will almost double to 70 million by 2030, therefore identifying therapeutic strategies for treating or preventing age-related disorders in humans is of major biomedical importance. Cardiovascular aging, defined as a reduction in vascular and cardiac functions with normal aging, occurs even in the absence of CVD risk factors and overt CVD. A key feature of cardiovascular aging is stiffening of the large elastic central arteries such as the aorta. This is important because aortic stiffness directly contributes to clinical problems such as increased blood pressure, reduced blood flow to the heart muscle, and thickening of the heart muscle. Therefore, these clinical consequences are hypothesized to mediate a substantial proportion of the increase in CVD risk in older adults. However, effective drug treatments for aortic stiffness are not currently available and the biological reasons (mechanisms) involved in causing aortic stiffening remain undefined. In addition, the inability of smaller blood vessels to relax, impairment of the heart to relax during the filling phase of the heart cycle (i.e., diastole), and increased blood pressure variability, have all been linked to aortic stiffness. Furthermore, chronic low-grade inflammation with advancing age has been proposed to be a common mechanistic link (i.e., biological reason) between these reductions in cardiovascular function in older adults. Therefore, the investigators propose that inflammation could be a novel therapeutic target to treat cardiovascular aging in older adults. Our central hypothesis is that inflammation mediates the age-related deterioration in cardiovascular functions observed with advancing age through the development of oxidative stress (i.e., imbalance between damaging oxygen free radicals vs. protective antioxidants). Our hypothesis predicts that chronic inhibition of inflammation with Salsalate, an FDA-approved anti-inflammatory drug similar to aspirin that is used to treat rheumatoid arthritis pain and known to inhibit the 'master' regulator of inflammation in the cell (i.e., nuclear factor kappa B), will improve cardiovascular function in older adults. In addition, the investigators hypothesize that the mechanism for the improvement in cardiovascular function during inhibition of inflammation will be by suppressing oxidative stress. To test our hypothesis, the investigators will randomize older healthy adults (age 50-79 years) to 3 g/day of salsalate or placebo (i.e., pill with inactive substance) pills for 4 weeks and have cardiovascular function measured at baseline and again after 4 weeks.

DETAILED DESCRIPTION:
Aim 1: To measure aortic wall stiffness and circulating biomarkers of oxidative stress during both acute (IV) intravenous infusions of saline and then the antioxidant vitamin C at baseline and after 4 weeks of salsalate or placebo in healthy older adults. Hypothesis 1: Inhibition of inflammation in older adults will decrease aortic wall stiffness in part by reductions in oxidative stress.

Aim 2: To measure brachial artery endothelium-dependent vasodilation (EDV) and circulating markers of oxidative stress during acute intravenous infusions of saline and then the vitamin C at baseline and after 4 weeks of salsalate or placebo in healthy older adults. Hypothesis 2: Inhibition of inflammation in older adults will improve vascular endothelial vasodilatory function in older adults in part by reductions in oxidative stress.

Aim 3: To measure left ventricular (LV) diastolic relaxation and filling dynamics and circulating markers of oxidative stress during both acute intravenous infusions of saline and then vitamin C at baseline and after 4 weeks of Salsalate or placebo in healthy older adults. Hypothesis 3: Inhibition of inflammation in older adults will improve LV diastolic function in part by reductions in oxidative stress.

Exploratory Aim: To measure 24-hour pressure variability and short-term baroreflex sensitivity before and after 4 weeks of oral Salsalate or placebo treatment in older adults. Exploratory hypothesis: Inhibition of inflammation in older adults will improve cardiovascular autonomic dysregulation in older healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 50 and < or = 79 years (older) or > or = 18 and < or = 39 years of age
* healthy, as determined by health history questionnaire, medical history and physical examination by physician or nurse practitioner, blood and urine chemistries, resting blood pressure and exercise 12-lead ECG
* blood chemistries indicative of normal renal (creatinine <2.2 mg/dl), normal liver, i.e., <3 times upper limit for alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and thyroid function (TSH between 0.4 - 5.0 mU/L)
* If currently receiving treatment with or taking any of the following supplements, be willing and able to discontinue taking them for 2 weeks prior and throughout the treatment period: Vitamin C, E or other multivitamins containing vitamin C or E; nutraceuticals containing vitamin C or E
* No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), Type 2 diabetes, chronic obstructive pulmonary or peripheral arterial disease
* Middle-aged/older females will be postmenopausal at least 1 year, had tubal ligation at least 1 year prior to screening, or who have had a total hysterectomy.
* Sedentary or recreationally active defined as performs regular aerobic exercise (30 min or more of vigorous walking, jogging, swimming, cycling, etc) less than 3 days/week or less than 12 days/month over the last year
* Non-smokers, defined as no history of smoking, no smoking for at least the past 1 year
* Normal resting 12-lead ECG.

Exclusion Criteria:

* History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, Type 2 diabetes and Type 1 diabetes
* Smoking or history of smoking within past one year
* History of gastric ulcers, bleeding disorders, dyspepsia, severe gastroesophageal reflux disease (GERD), or metabolic acidosis
* History of asthma or lung disease (chronic obstructive pulmonary disease, COPD)
* Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree atrioventricular (AV) block, atrial fibrillation/flutter)
* Serious neurologic disorders including seizures
* History of renal failure, dialysis or kidney transplant
* Serum creatinine > 2.2 mg/dL, or hepatic enzyme concentrations > 3 times the upper limit of normal
* History of HIV infection, hepatic cirrhosis, other preexisting liver disease, or positive HIV, Hepatitis B or C test at screening.
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* History of recent chicken pox, shingles or influenza (ie., risk of Reye's syndrome) Recent flu-like symptoms within the past 2 weeks
* Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.
* Women with history of hormone replacement therapy within the past 6 months
* History of rheumatoid arthritis, Grave's disease, systemic lupus erythematosis, and Wegener's granulomatosis;
* Taking medications for diabetes mellitus, kidney disease, liver disease, asthma, sepsis or seizure disorders;
* Taking lipid lowering (e.g., statins, niacin), glycemic control (e.g. metformin, insulin), anticoagulation, anti-seizure, anti-depression or antipsychotic agents
* History of co-morbid condition that would limit life expectancy to < 6 months.
* It is unknown if Salsalate is transferred in seminal fluid of men. However, it is recommended that proper protection such as a condom be used during intercourse during the study.
* Concomitant treatment with: aspirin, baby aspirin, indomethacin, naproxen (Aleve), acetaminophen (Tylenol), ibuprofen (Advil, Motrin), any other non-steroidal anti-inflammatory drugs; cox-2 inhibitors (Celebrex, Vioxx, etc); allopurinol (Zyloprim, Lopurin, Allopurin; coumadin (Warfarin), enoxaparin (Lovenox); clopidogrel (Plavix); dipyridamole (Persantine); heparin; diabetic medications (Metformin, glyburide, insulin, etc), thiazolidinediones (Avandia, Rezulin, Actos); corticosteroids (prednisone); methotrexate, infliximab (Remicade), etanercept (Enbrel); levothyroxine (Levoxyl, Synthroid, Levoxyl, Unithroid); Levodopa; Phosphodiesterase (PDE) 5 inhibitors (e.g., Viagra®, Cialis®, Levitra®, or Revatio®); PDE 3 inhibitors (e.g., cilostazol, milrinone, or vesnarinone); lithium
* May participate if use of the following medications are discontinued 2 weeks prior to participation: salicylate medications, aspirin, antioxidants, herbal supplements, vitamins, omega-3 fatty acids; cox-2 inhibitors (Celebrex, Vioxx, etc)
* May participate if no use of the following medications in the 48 hours prior to experimental visits: naproxen (Aleve), acetaminophen (Tylenol), ibuprofen (Advil, Motrin), other any non-steroidal anti-inflammatory drugs
* Vulnerable populations (prisoners, etc.) are not included in this study because we are studying healthy middle-aged/older adults.
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
* Hemoglobin <12 mg/dl for men; < 10 mg/dl for women
* History of alcohol abuse or >10 alcoholic units per week (1 unit= 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 oz alcohol)
* Low platelets (<100,000 cu mm)
* On weight loss drugs (e.g., Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanol-amine), or similar over-the-counter medications) within 3 months of screening
* Any surgery within 30 days of screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Pyle L, Staten MA, Shoelson SE; TINSAL-T2D (Targeting Inflammation Using Salsalate in Type 2 Diabetes) Study Team. The effects of salsalate on glycemic control in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2010 Mar 16;152(6):346-57. doi: 10.7326/0003-4819-152-6-201003160-00004. PMID 20231565
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Jablonski KL, Chonchol M, Pierce GL, Walker AE, Seals DR. 25-Hydroxyvitamin D deficiency is associated with inflammation-linked vascular endothelial dysfunction in middle-aged and older adults. Hypertension. 2011 Jan;57(1):63-9. doi: 10.1161/HYPERTENSIONAHA.110.160929. Epub 2010 Nov 29. PMID 21115878
- [Background] McCarty MF. Salsalate may have broad utility in the prevention and treatment of vascular disorders and the metabolic syndrome. Med Hypotheses. 2010 Sep;75(3):276-81. doi: 10.1016/j.mehy.2009.12.027. Epub 2010 Jan 18. PMID 20080359
- [Background] Pierce GL, Lesniewski LA, Lawson BR, Beske SD, Seals DR. Nuclear factor-kappaB activation contributes to vascular endothelial dysfunction via oxidative stress in overweight/obese middle-aged and older humans. Circulation. 2009 Mar 10;119(9):1284-92. doi: 10.1161/CIRCULATIONAHA.108.804294. Epub 2009 Feb 23. PMID 19237660
- [Background] Lesniewski LA, Durrant JR, Connell ML, Folian BJ, Donato AJ, Seals DR. Salicylate treatment improves age-associated vascular endothelial dysfunction: potential role of nuclear factor kappaB and forkhead Box O phosphorylation. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):409-18. doi: 10.1093/gerona/glq233. Epub 2011 Feb 8. PMID 21303813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 59 participants were consented/enrolled. A total of 13 were excluded or lost to follow up after consent (n=8 did not meet inclusion criteria after screening; n=1 lost to follow up; n=1 time committment; n=1 moved out of state; n=2 other).
Groups:
- Salsalate: Salsalate capsule 1.5 g twice per day by mouth for 4 weeks
  Salsalate
- Placebo: Placebo capsule twice per day by mouth for 4 weeks
  Placebo (for salsalate)
- Young Control: No intervention; Baseline measurements only, participants not randomized
Period: Overall Study
Arm/Group | Salsalate | Placebo | Young Control
Started | 14 | 14 | 17
Completed | 11 | 13 | 17
Not Completed | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Salsalate: Salsalate capusule 1.5 g twice per day by mouth for 4 weeks
- Young Control: No intervention, not randomized; Baseline measurements only
- Total: Total of all reporting groups
Arm/Group | Salsalate | Placebo | Young Control | Total
Number analyzed (Participants) | 14 | 14 | 17 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (7.4) | 55.8 (5.3) | 26.2 (5.2) | 48.1 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 7 | 24
  Male | 6 | 5 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Carotid-femoral Pulse Wave Velocity (CFPWV)
Description: Aortic stiffness
Time Frame: Change in CFPWV from baseline at 4 weeks
Population: After baseline measurements, there were 3 dropouts in salsalate group for a total of 11 completed in salsalate, and 1 dropout in the placebo group for a total of 13 completed in placebo.
Measure: Mean (Standard Error); unit: cm/sec
Groups:
- Salsalate: Received 4 weeks of daily oral salsalate
- Placebo: Received 4 weeks of placebo
- Young Control Group: No Intervention; Baseline measurements only, participants not randomized
Arm/Group | Salsalate | Placebo | Young Control Group
Number analyzed (Participants) | 14 | 14 | 17
cm/sec
  Baseline | 831.3 (45.3) | 785.1 (41.1) | 538.0 (17.9)
  4 weeks: number analyzed (Participants) | 11 | 13 | 17
  4 weeks | 839.6 (66.4) | 740.01 (45.6) | NA (NA) — Data not collected from any participant in the Young Control Arm/Group at 4 weeks

2. Secondary Outcome: Brachial Artery Flow-mediated Dilation (FMD)
Description: Endothelial function
Time Frame: Change from baseline brachial artery FMD at 4 weeks
Population: After baseline measurements, there were 3 dropouts in salsalate group and 1 FMD that was not able to be anayzed (poor image quality) for a total of 10 in salsalate for FMD. There was 1 dropout in the placebo group and 2 FMDs not analyzed (poor image quality) for a total of 11 analyzed in placebo for FMD.
Measure: Mean (Standard Error); unit: Percent dilation
Groups:
- Salsalate: Salsalate capsule 1.5 g twice per day by mouth for 4 weeks
- Young Control Group: No intervention; Baseline measurements only; participants not randomized
Arm/Group | Salsalate | Placebo | Young Control Group
Number analyzed (Participants) | 14 | 14 | 17
Percent dilation
  Baseline: number analyzed (Participants) | 14 | 12 | 17
  Baseline | 3.49 (1.05) | 3.57 (1.14) | 5.88 (0.97)
  4 Weeks: number analyzed (Participants) | 10 | 11 | 17
  4 Weeks | 4.60 (1.24) | 2.50 (1.32) | NA (NA) — Only baseline date were collected, no 4 week data were collected.

3. Other Pre Specified Outcome: Tissue Doppler Left Ventricular Relaxation Velocity (E')
Description: Left ventricular diastolic dysfunction
Time Frame: Change from baseline E' at 4 weeks
Population: Data were not obtained because cardiac echos could not be performed in participants because of lack of equipment
Groups:
- Placebo: Placebo capsules twice per day by mouth for 4 weeks
Arm/Group | Salsalate | Placebo | Young Control Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Salsalate: Salsalate 1.5 g twice per day by mouth for 4 weeks
- Placebo: Placebo capusule twice per day by mouth for 4 weeks
Arm/Group | Salsalate | Placebo | Young Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=14) | Placebo (N=14) | Young Control Group (N=17)
Elevated AST/ALT (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — Elevated serum AST/ALT after 2 weeks of salsalate that resolved within 7 days after stopping medications without complication
Allergic reaction (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — One participant in placebo group developed allergic reaction (facial / orbital swelling) but after withdrawl from study and PI unblinded it was determined that the participant was in the placebo group. Follow up likley allergy to shellfish.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes